CLINICAL TRIAL: NCT00343577
Title: Observational Study of Antiproteinuric Agents in Patients With Fabry Disease Treated With Enzyme Replacement Therapy
Brief Title: Antiproteinuric Agents and Fabry Disease
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Other Study IDs: X050202007
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2006-06

CONDITIONS: Fabry Disease; Proteinuria
Keywords: proteinuria; ARBs; agalsidase-beta; MDRD estimated GFR; Chronic kidney disease
MeSH Terms: conditions — Fabry Disease; Proteinuria; Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Fabry disease is a rare disorder that often has kidney involvement with increased urine protein excretion. Proteinuria is recognized as an important risk factor for progression of chronic kidney disease. Our hypothesis is that using drugs that reduce urine protein excretion (ACE inhibitors and ARBs) will have a beneficial effect on patients with Fabry disease who already are receiving enzyme replacement therapy. A longitudinal, observational study is being undertaken to determine the utility of these agents in Fabry disease, realizing that these agents are primarily indicated for reducing systemic blood pressure, and most patients with Fabry disease have relatively low blood pressures at baseline.

DETAILED DESCRIPTION:
Fabry disease is a rare disorder that often has kidney involvement with increased urine protein excretion. Proteinuria is recognized as an important risk factor for progression of chronic kidney disease. Our hypothesis is that using drugs that reduce urine protein excretion (ACE inhibitors and ARBs) will have a beneficial effect on patients with Fabry disease who already are receiving enzyme replacement therapy. A longitudinal, observational study is being undertaken to determine the utility of these agents in Fabry disease, realizing that these agents are primarily indicated for reducing systemic blood pressure, and most patients with Fabry disease have relatively low blood pressures at baseline.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed Fabry disease
* institution of commercially available agalsidase-beta

Exclusion Criteria:

* s/p kidney transplant

Ages: 14 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2001-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: David G Warnock, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Tahir H, Jackson LL, Warnock DG. Antiproteinuric therapy and fabry nephropathy: sustained reduction of proteinuria in patients receiving enzyme replacement therapy with agalsidase-beta. J Am Soc Nephrol. 2007 Sep;18(9):2609-17. doi: 10.1681/ASN.2006121400. Epub 2007 Jul 26. PMID 17656478